CLINICAL TRIAL: NCT02993926
Title: An Observational, Retrospective Study to Evaluate the Long Term Safety and Effectiveness of Leuprorelin in the Treatment of Central Precocious Puberty
Brief Title: A Study to Assess the Safety and Efficacy of Enantone (Leuprorelin) in Central Precocious Puberty (CPP) Among Chinese Participants
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Leuprorelin-5001
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Central Precocious Puberty
Keywords: Drug Therapy
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment Phase: Enantone: Participants with CPP who were treated with Enantone (≥ 30 μg/kg up to 180 μg/kg) for at least 9 continuous months and who initiated and received the last dose of treatment during the index period from 01 September 1998 to 30 September 2018 (the mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months).
  Interventions: Drug: Enantone
- Follow Up: Participants No longer Treated for CPP: Participants who had completed their CPP during the treatment phase with Enantone and were no longer on treatment in the follow-up phase (the mean duration of follow up was 8.75 months with a range of 1.9 to 29.5 months).
- Follow Up: Treated with Non-Enantone GnRHa after Enantone: Participants who were continuing their CPP treatment with a non-Enantone gonadotropin releasing hormone agonist (GnRHa) after treatment with Enantone in the follow-up phase (the mean duration of follow up while on another GnRHa was 10.80 months with a range of 2.8 to 20.5 months, and the mean duration of follow up after stopping treatment was 4.26 months with a range of 0.0 [i.e. 1 day] to 12 months).
  Interventions: Drug: GnRH agonist

INTERVENTIONS:
Drug: Enantone — Enantone suspension for injection
  Other Names: Leuprorelin
  Groups: Treatment Phase: Enantone
Drug: GnRH agonist — A non-Enantone GnRH agonist
  Groups: Follow Up: Treated with Non-Enantone GnRHa after Enantone

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of Enantone in the treatment of CPP in Chinese participants.

DETAILED DESCRIPTION:
The drug being evaluated in this study is called Enantone (leuprorelin). Enantone is used to treat children who have CPP. This study will look at long term safety and efficacy of leuprorelin in the treatment of Chinese participants with CPP.

The study will enroll approximately 300 participants.

All participants who have received leuprorelin 30 mcg/kg to <90 mcg/kg or 90 mcg/kg to 180 mcg/kg per body weight, injection, subcutaneously, every 4 weeks up to at least 9 continuous months during the index period from September 1st 1998 to September 30th 2018 will be observed.

This multi-center trial will be conducted in China. Data will be collected over period of 20 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has diagnosis of idiopathic CPP.
2. Has been treated with leuprorelin acetate (Enantone) for at least 9 continuous months of therapy with either a stable dose of high dose (greater than or equal to [>=] 90 mcg/kg up to 180 mcg/kg) or low dose (< 90 mcg/kg down to 30 mcg/kg).
3. Has initiated and completed treatment during the index period from September 1st 1998 to September 30th 2018.
4. Have the following information prior to initiation of enantone and at least one record of each of the following parameters at the end of enantone treatment in the medical records: Tanner staging, estradiol or testosterone level, and FSH and LH level. The participant should have at least one record of bone age prior to the initiation gonadotropin releasing hormone analogs (GnRHa) therapy with enantone to support the diagnosis of CPP. In addition, should have at least one record of bone age during treatment with enantone.

Exclusion Criteria:

1. Has been treated with leuprorelin acetate or any other GnRHa for conditions other than CPP.
2. Has used any other GnRHa products for CPP treatment prior to initiation of enantone therapy.
3. CPP participants with identified etiology, such as brain tumor or cranial irradiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with CPP will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-06-24 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (6):
- China (6):
  - The Children's Hospital, Zhejiang University School of Medicine, Wuhan, Hubei
  - Childrens Hospital of Hunan province, Changsha, Hunan
  - Jiangsu Province Hosptial, Nanjing, Jiangsu
  - Children's Hospital of Jiangxi province, Nanchang, Jiangxi
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in China from 24 Jun 2017 to 30 Sep 2018.
Pre-assignment Details: Participants with a diagnosis of central precocious puberty (CPP) who previously received Enantone for at least 9 continuous months in clinical practice index period: 1 September 1998 to 30 September 2018 were enrolled in this study.
Period: Enantone Treatment Phase
Arm/Group | Treatment Phase: Enantone | Follow Up: Participants No Longer Treated for CPP | Follow Up: Treated With Non-Enantone GnRHa After Enantone
Started | 108 | 0 | 0
Completed | 76 | 0 | 0
Not Completed | 32 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Changed CPP Therapy to Another GnRHa | 26 | 0 | 0
Not completed — Investigator Judgment | 1 | 0 | 0
Not completed — Reason Not Specified | 4 | 0 | 0
Period: Follow-Up Phase
Arm/Group | Treatment Phase: Enantone | Follow Up: Participants No Longer Treated for CPP | Follow Up: Treated With Non-Enantone GnRHa After Enantone
Started | 0 | 44 | 26
Completed | 0 | 44 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled participants.
Arm/Group | Treatment Phase: Enantone
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] — Age presented here is age at enantone treatment initiation (Years).
  years | 8.45 (1.124)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 108
Tanner Staging Evaluation [Count of Participants; unit: Participants] — Tanner Stage is used to define physical measurements of sexual development based on external primary and secondary sex characteristics. Female and male participants were evaluated for breast development and genital development respectively and both genders for pubic hair distribution based on a 5-stage scale ranging from Stage I (prepubertal/preadolescent characteristics) to Stage V (mature or adult characteristics). Participants classified as having progression if either breast/genitals or pubic hair were present. Otherwise participant is classified as regression or no progression.
  Participants
    Breast (Female) and Genitals (Male), Stage I | 1
    Breast (Female) and Genitals (Male), Stage II | 49
    Breast (Female) and Genitals (Male), Stage III | 46
    Breast (Female) and Genitals (Male), Stage IV | 3
    Pubic Hair, Stage I | 75
    Pubic Hair, Stage II | 14
Peak Stimulated Luteinizing Hormone (LH) [Mean (Standard Deviation); unit: U/L] | 16.935 (10.7717)
Peak Stimulated Follicle Stimulating Hormone (FSH) [Mean (Standard Deviation); unit: U/L] | 14.407 (5.9366)
Estradiol [Mean (Standard Deviation); unit: ng/L] | 23.3453 (18.1633)
Testosterone [Mean (Standard Deviation); unit: pg/mL] | 70.4653 (127.7357)
Bone Age/Chronological Age Ratio [Mean (Standard Deviation); unit: ratio] — Bone age (BA) was estimated using an X-ray. Chronological age (CA) at the date of corresponding X-ray (Date of X-ray - Date of birth)/365.25. Ratio of BA/CA was calculated.
  ratio | 1.22 (0.122)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE) During Enantone Treatment Phase
Description: A TEAE is any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: During treatment with and up to 30 days post last dose of Enantone (the mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months)
Population: Safety Analysis Set included all enrolled participants. Data in this outcome measure is reported separately for male and female participants.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Phase: Enantone (Male): Male participants with CPP who were treated with Enantone (≥ 30 μg/kg up to 180 μg/kg) for at least 9 continuous months and who initiated and received the last dose of treatment during the index period from 01 September 1998 to 30 September 2018 (the mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months).
- Treatment Phase: Enantone (Female): Female participants with CPP who were treated with Enantone (≥ 30 μg/kg up to 180 μg/kg) for at least 9 continuous months and who initiated and received the last dose of treatment during the index period from 01 September 1998 to 30 September 2018 (the mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months).
Arm/Group | Treatment Phase: Enantone (Male) | Treatment Phase: Enantone (Female)
Number analyzed (Participants) | 4 | 104
Participants
  TEAE | 4 | 71
  SAE | 0 | 2

2. Primary Outcome: Number of Participants With at Least One Treatment Emergent Adverse (TEAE) and Serious Adverse Event (SAE) During Follow-up Phase
Description: as for outcome 1
Time Frame: Mean duration of follow-up=8.75 months (range: 1.9-29.5 months) for No longer treated for CPP group; 10.80 months (range: 2.8-20.5 months) for Treated with Non-Enantone GnRHa group after treatment with Enantone (while on another GnRHa)
Population: Safety Analysis Set included all enrolled participants. Data in this outcome measure is reported separately for male and female participants for follow-up period. There were no observations available for male participants who continued therapy with a Non-Enantone GnRHa in the follow-up period.
Measure: Count of Participants; unit: Participants
Groups:
- Follow UP: Participants No Longer Treated for CPP (Male): Male participants who had completed their CPP during the treatment phase with Enantone and were no longer on treatment in the follow-up phase (the mean duration of follow up was 8.75 months with a range of 1.9 to 29.5 months).
- Follow Up: Participants No Longer Treated for CPP (Female): Female participants who had completed their CPP during the treatment phase with Enantone and were no longer on treatment in the follow-up phase (the mean duration of follow up was 8.75 months with a range of 1.9 to 29.5 months).
- FollowUp:Treated With Non-Enantone GnRHa After Enantone-Female: Female participants who were continuing their CPP treatment with a non-Enantone GnRHa after treatment with Enantone in the follow-up phase (the mean duration of follow up while on another GnRHa was 10.80 months with a range of 2.8 to 20.5 months, and the mean duration of follow up after stopping treatment was 4.26 months with a range of 0.0 [i.e. 1 day] to 12 months).
Arm/Group | Follow UP: Participants No Longer Treated for CPP (Male) | Follow Up: Participants No Longer Treated for CPP (Female) | FollowUp:Treated With Non-Enantone GnRHa After Enantone-Female
Number analyzed (Participants) | 2 | 42 | 26
Participants
  TEAE | 0 | 10 | 9
  SAE | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Had Regression or No Progression in Tanner Staging at the End of Enantone Treatment Phase
Description: Tanner Stage is used to measure pubertal development. Female (F) and male (M) participants were evaluated for breast development and genital development respectively and both genders for pubic hair development. Tanner Stage is based on progression through 5-stages. Participants were classified as having progression if either breast/genitals or pubic hair progression were present. Otherwise participant is classified as regression or no progression.
Time Frame: The mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months
Population: Full Analysis Set (FAS) included all enrolled participants. Number of participants analyzed is the number of male or female participants with data available for the analysis of this outcome measure at the end of Treatment Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Enantone (Male) | Treatment Phase: Enantone (Female)
Number analyzed (Participants) | 1 | 79
percentage of participants | 0 [0 to 97.50] | 79.7 [69.20 to 87.96]

4. Primary Outcome: Percentage of Participants Who Had Regression or No Progression in Tanner Staging at the End of Follow-Up Phase
Description: as for outcome 3
Time Frame: No longer treated for CPP group - Month: 27 (766- 855 days) post last dose of Enantone; Treated with Non-Enantone GnRHa group - Month 21 (586- 675 days) post last dose of Enantone
Population: FAS included all enrolled participants. Number of participants analyzed is the number of male or female participants with data available for analysis of this outcome measure at the end of Follow-up Phase. There were no observations available for male participants who continued therapy with a Non-Enantone GnRHa in the follow-up period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Follow UP: Participants No Longer Treated for CPP (Male) | Follow Up: Participants No Longer Treated for CPP (Female) | FollowUp:Treated With Non-Enantone GnRHa After Enantone-Female
Number analyzed (Participants) | 0 | 0 | 1
percentage of participants |  |  | 0 [0 to 97.5]

5. Secondary Outcome: Percentage of Participants With Post Stimulation Test Peak Values, for Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH), Suppressed Below Upper Limit Value (ULV) at the End of Enantone Treatment Phase
Description: The LH suppression is defined as peak LH ≤2 U/L for female and peak LH ≤2.7 U/L for male. The FSH suppression is defined as peak FSH ≤6.7 U/L for female and peak FSH ≤3.7 U/L for male. Post Stimulation Test, the peak values for LH and FSH suppression below Upper Limit Value (ULV) are reported.
Time Frame: The mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months
Population: FAS included all enrolled participants. Number of participants analyzed is the number of male or female participants with data available for analysis of this outcome measure at the end of Treatment Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Enantone (Male) | Treatment Phase: Enantone (Female)
Number analyzed (Participants) | 1 | 52
percentage of participants
  LH (U/L) Peak Value ≤ ULV | 100 [2.50 to 100] | 98.1 [89.74 to 99.95]
  FSH (U/L) Peak Value ≤ ULV | 100 [2.50 to 100] | 100 [93.15 to 100]

6. Secondary Outcome: Percentage of Participants With Post Stimulation Test Peak Values, for Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH), Suppressed Below Upper Limit Value (ULV) at the End of Follow-Up Phase
Description: as for outcome 5
Time Frame: as for outcome 4
Population: No data were available for this outcome measure.
Arm/Group | Follow UP: Participants No Longer Treated for CPP (Male) | Follow Up: Participants No Longer Treated for CPP (Female) | FollowUp:Treated With Non-Enantone GnRHa After Enantone-Female
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Value, for Estradiol or Testosterone, Suppressed Below Upper Limit Value (ULV) at the End of Enantone Treatment Phase
Description: Estradiol or Testosterone, suppressed below Upper Limit Value (ULV) were reported. The ULV for estradiol and testosterone were 20 pg/mL and 7.34 nmol/L, respectively.
Time Frame: The mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months
Population: FAS included all enrolled participants. Number of participants analyzed is the number of male or female participants with data available for analysis of this outcome measure at the end of Treatment Phase. There were no observations available for male participants who continued therapy with a Non-Enantone GnRHa in the follow-up period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Enantone (Male) | Treatment Phase: Enantone (Female)
Number analyzed (Participants) | 4 | 103
percentage of participants | 100 [39.76 to 100.00] | 74.8 [65.24 to 82.80]

8. Secondary Outcome: Percentage of Participants With Value, for Estradiol or Testosterone, Suppressed Below Upper Limit Value (ULV) at the End of Follow-Up Phase
Description: as for outcome 7
Time Frame: No longer treated for CPP group-Month: 27 (766-855 days) post last dose of Enantone; Treated with Non-Enantone GnRHa group-Month 21 (586-675 days) post last dose of Enantone
Population: FAS included all enrolled participants. Number of participants analyzed is the number of male or female participants with data available for analysis of analysis at the end of Follow-up Phase. There were no observations available for male participants who continued therapy with a Non-Enantone GnRHa in the follow-up period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Follow UP: Participants No Longer Treated for CPP (Male) | Follow Up: Participants No Longer Treated for CPP (Female) | FollowUp:Treated With Non-Enantone GnRHa After Enantone-Female
Number analyzed (Participants) | 0 | 1 | 1
percentage of participants |  | 0 [0 to 97.5] | 0 [0 to 97.5]

9. Secondary Outcome: Percentage of Participants With Decease of Ratio of Bone Age to Chronological Age at the End of Enantone Treatment Phase
Description: Bone age (BA) was estimated using an X-ray. Chronological age (CA) at the date of corresponding X-ray (Date of X-ray - Date of birth)/365.25. Ratio of BA/CA was calculated.
Time Frame: The mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Enantone (Male) | Treatment Phase: Enantone (Female)
Number analyzed (Participants) | 4 | 92
percentage of participants | 75.0 [19.41 to 99.37] | 90.2 [82.24 to 95.43]

10. Secondary Outcome: Percentage of Participants With Decease of Ratio of Bone Age to Chronological Age at the End of Follow-up Phase
Description: as for outcome 9
Time Frame: No longer treated for CPP group - Month: 27 (766- 855 days) post last dose of Enantone; Treated with Non-Enantone GnRHa group - Month 18 (496-585 days) post last dose of Enantone
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Follow UP: Participants No Longer Treated for CPP (Male) | Follow Up: Participants No Longer Treated for CPP (Female) | FollowUp:Treated With Non-Enantone GnRHa After Enantone-Female
Number analyzed (Participants) | 0 | 2 | 3
percentage of participants |  | 100 [15.81 to 100] | 100 [29.24 to 100]

ADVERSE EVENTS:
Time Frame: Treatment Phase - During treatment with Enantone and up to 30 days post last dose of Enantone (mean duration of Enantone exposure was 22.3 months, ranging from 10.1 to 52.4 months); Follow-up Phase: No Longer Treated for CPP group - mean duration of follow up was 8.75 months with a range of 1.9 to 29.5 months; Treated with Non-Enantone GnRHa group - mean duration of follow up while on another GnRHa was 10.80 months with a range of 2.8 to 20.5 months.
Arm/Group | Treatment Phase: Enantone | Follow Up: Participants No Longer Treated for CPP | Follow Up: Treated With Non-Enantone GnRHa After Enantone
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/44 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/108 | 0/44 | 0/26
Other Adverse Events (participants affected / at risk) | 63/108 | 0/44 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: Enantone (N=108) | Follow Up: Participants No Longer Treated for CPP (N=44) | Follow Up: Treated With Non-Enantone GnRHa After Enantone (N=26)
Pneumonia (Infections and infestations) | 1 | 0 | 0
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: Enantone (N=108) | Follow Up: Participants No Longer Treated for CPP (N=44) | Follow Up: Treated With Non-Enantone GnRHa After Enantone (N=26)
Upper respiratory tract infection (Infections and infestations) | 18 | 0 | 1
Growth retardation (Musculoskeletal and connective tissue disorders) | 15 | 0 | 2
Bronchitis (Infections and infestations) | 14 | 0 | 0
Pharyngitis (Infections and infestations) | 13 | 0 | 1
Pyrexia (General disorders) | 9 | 0 | 2
Refraction disorder (Eye disorders) | 9 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2
Rhinitis (Infections and infestations) | 7 | 0 | 0
Tonsillitis (Infections and infestations) | 7 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 0 | 0
Bone density decreased (Investigations) | 4 | 0 | 0
Conjunctivitis (Infections and infestations) | 4 | 0 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Growth hormone deficiency (Endocrine disorders) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Immunodeficiency (Immune system disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Keratosis follicular (Congenital, familial and genetic disorders) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vulvitis (Infections and infestations) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The enrollment of only 100 participants did not support the performance of subgroup analysis of outcomes by dose. Retrospective observational data is not controlled and therefore robust analysis could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications and presentations must be prepared in accordance with this section and the Clinical Study Site Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT02993926/Prot_001.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02993926/SAP_000.pdf